CLINICAL TRIAL: NCT06771505
Title: SBS DISK- Creation of a Quality of Life Tool for Short Bowel Patients Compared With a Validated Quality of Life Questionnaire (SBS QoL)
Acronym: SBS DISK
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0889; 2024-A02032-45 (Other: ID-RCB)
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Short Bowel Syndrome
Keywords: Short Bowel syndrome; Quality of life
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire completion: The partient completes the two quality of life assessment questionnaires (Short Bowel Syndrome Quality of Life (SBS QoL) and SBS disk assessment tool), in paper format.

SUMMARY:
Patients with short bowel syndrome have an impact on their quality of life because they need temporary or permanent parenteral nutritional support. The quality of life of these patients has been the subject of several studies and assessment tools exist, such as the Short Bowel Syndrome Quality of Life (SBS QoL). This tool may seem complex and tedious to use in everyday practice. However, it is important to regularly assess the quality of life of these patients. This is why the investigators are proposing to create a new tool for more rapid assessment of the quality of life of patients with short bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Patient able to read and speak French
* Patient suffering from short bowel syndrome

Exclusion Criteria:

* Known cognitive disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will focus on adult patients with short bowel syndrome followed up in the GHS Intensive Clinical Nutrition Department, during a consultation, a day hospital or a conventional hospital stay.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Validation of a new quality of life tool, the SBS disk, in comparison with a quality of life assessment tool, the SBS QoL. | Day 1
  Self-questionnaire in the form of a disk which covers 10 themes: Energy, stress level, anxiety, diet, abdominal pain, transit, appliances, social life, social and professional activity, sleep, as well as self-image and intimate life, according to the recommendations of the WHO quality of life assessment.
  These themes are the same as those generally covered by the SBS QoL reference questionnaire, with the exception of self-image and intimacy.
  The themes are evaluated according to the patient's feelings during the past week on a scale from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte BERGOIN, Doctor, Principal Investigator — Service d'hépato-gastro-entérologie et Assistance nutritionnelle - Hôpital Lyon Sud - CHLS
Locations (1):
- Hôpital Lyon Sud - CHLS, Pierre-Bénite, France